CLINICAL TRIAL: NCT01360060
Title: Analgesia After Cesarean Section
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Hyoseok, Na/professor, Seoul National University Bundang Hospital
Other Study IDs: Mg_section
Record Dates: First submitted 2011-05-17; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Preeclampsia; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Group N: parturients who had undergone Cesarean section under the diagnosis of non-preeclampsia
- Group P: parturients who had undergone Cesarean section under the diagnosis of preeclampsia
  Interventions: Drug: Magnesium Sulphate

INTERVENTIONS:
Drug: Magnesium Sulphate — Magnesium sulphate was infused for the management of preeclampsia at perioperative period.
  Groups: Group P

SUMMARY:
Magnesium sulphate is the first line therapy for the management of preeclampsia and eclampsia in obstetrics. Perioperative administration of magnesium sulphate has been proved to be an effective as an analgesic adjuvant. The investigators evaluated the analgesic effect of magnesium in parturients undergoing Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* parturients undergoing Cesarean section

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: medical record review
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change of numeric rating scale (NRS) of postoperative pain during postoperative period | postoperative 1, 2, 3, and 4 day

SECONDARY OUTCOMES:
incidence of stopping of intravenous PCA during postoperative 4 days | during postoperative 4 days
serum magnesium level of group P | preoperative 1 h and postoperative 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Gyeonggi-do, South Korea